CLINICAL TRIAL: NCT01252550
Title: Association Between GI Microbiota, Low-grade Inflammation and Classical Pathophysiological Factors in Patients With Irritable Bowel Syndrome (IBS) and Effect of the Consumption of Activia on GI Symptoms Provoked by a Lactulose Challenge Test in IBS Patients
Brief Title: Effects of Activia in IBS
Acronym: MOSAIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Principal Investigator, Magnus Simrén, Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NU341
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; GI; QOL; Pathophysiology; Gut microbiota; Danone; Activia; Probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Activia® (Active Comparator): Activia® (125g/pot)
  Interventions: Dietary Supplement: Activia® (125g/pot)
- Acidified non-fermented dairy product (Placebo Comparator): Acidified non-fermented dairy product (125g/pot)
  Interventions: Dietary Supplement: Acidified non-fermented dairy product

INTERVENTIONS:
Dietary Supplement: Activia® (125g/pot) — Activia® (125g/pot) - dairy product containing bacterial culture Acti Regularis®
  Arms: Activia®
Dietary Supplement: Acidified non-fermented dairy product — Acidified non-fermented dairy product (125g/pot)
  Arms: Acidified non-fermented dairy product

SUMMARY:
The purpose of this study is to investigate the association between gut microbiota, immunology and typical pathophysiological factors in patients with IBS (all subtypes) AND to assess the effect of Activia consumption on GI symptoms provoked by a lactulose challenge test in IBS patients.

DETAILED DESCRIPTION:
BACKGROUND

There is a wide variety of symptoms in IBS, irritable bowel syndrome, both among individuals and in the symptoms of a specific individual. Pathophysiological factors that are of importance have been identified in IBS, but all of the factors do not occur in the symptomatology of all patients. Visceral hypersensitivity, deviant motor and secretion function in the gastrointestinal tract as well as psychological factors are believed to be of importance. However the relative importance of specific factors in the symptomatology is not elucidated.

Deviations in the autonomic and central nerve function have also been demonstrated in IBS, along with low grad inflammation, immunological anomalies, and changes in the microbiological gut flora. The importance of these factors in developing the more established pathophysiological factors, visceral hypersensitivity, and deviated gastrointestinal motor and secretion functions have not yet been studied. Neither have the interactions between the autonomic and central nerve functions or the significance of these functions in IBS.

In response to the recent findings, regarding deviant microbiological gut flora in IBS, the use of probiotics as treatment has been tested, with altering outcome. The effects of some products are positive, but far from all the patients with IBS get sufficient relief. The response of treatment with probiotics cannot be predicted with the methods available today; in example it is not possible to predict which patient will respond to the treatment and what the mechanisms behind the symptom relief are.

Questions

* What affects the symptomatology in IBS?

  * Visceral hypersensitivity
  * Deviant colonic motor function
  * Autonomic nerve dysfunction
  * Central nerve dysfunction (especially in the level of the brain stem)
  * Psychological factors
  * Coping
  * Demography (sex, age)
  * Immunological deviations in peripheral blood/intestine
  * Deviations in the composition of the microbiological gut flora
  * Sexual/physical abuse
* What are the interactions between pathophysiological deviations in IBS?
* Can the treatment response of probiotics be predicted?
* Why do probiotics give relief to some of the patients with IBS?

INVESTIGATION

1. A structured investigational model, covering the most important pathophysiological factors in IBS and clarifying the symptomatology of the patients in detail.
2. A randomized, double blinded placebo controlled study, evaluating the effects of probiotics (Bifidobacterium lactis) on the symptomatology in IBS as well as measuring the effect probiotics have on the fermentation in the intestines, immunological variables and the composition of the microbiological gut flora.

VISIT 1

* The patients are thoroughly informed regarding the context of the study and a written consent is signed.
* Blood samples are taken to rule out any organic disease (Hb, LPK, TPK, Na, K, Crea, Liver status, CRP, Transglutaminase antibodies).
* Validated questionnaires are completed

  * IBS Symptom Severity Scale (IBS-SSS) - gastrointestinal and extra intestinal symptoms
  * Gastrointestinal Symptom Rating Scale - IBS (GSRS-IBS) - IBS specific GI-symptoms
  * Hospital Anxiety and Depression Scale (HAD) - general anxiety and depression
  * Visceral Sensitivity Index (VSI) - GI-specific anxiety
  * Patient Health Questionnaire-15 (PHQ-15) - severity of somatisation, depression, anxiety (panic anxiety, eating disorders and alcohol problems)
  * IBS Quality of Life Questionnaire (IBSQOL) - disease specific health related quality of life
  * Fatigue Impact Scale (FIS) - impact of fatigue on quality of life
  * Abuse Questionnaire - physical and sexual abuse
  * Sense of Coherence Index - sense of coherence, coping
* ABR (Auditory Brain stem Response audiometry) - brain stem audiometry measuring the electric activity in level of the brain stem while listening to different audio stimuli (listening to sounds of clicks through headphones). Through this test the function of the brain stem can be measured, its ability to mask the effect of disturbing noises etc.
* Holter-ECG (24 h) - spectrum analysis to evaluate the autonomic nerve function; the balance between parasympathetic and sympathetic nerve function.
* Permeability test of the intestine - the patient drinks a liquid solution of water and sugars (50.0 g sucrose, 5.0 g mannitol, 10.0 g lactulose and 1.0 g sucralose in 200 ml tap water), thereafter urine is collected during the following 9 h. The amount of sugars found in the urine is a measurement of the permeability in the intestines. The urine will be collected in separate containers depending on what time of the day it is, and depending on the time the permeability in the small intestine respectively in the large intestine can be measured separately.
* Registration of stool consistency and frequency over the following 2-3 weeks, until visit 3, using the "Bristol Stool Form Scale" (BSF)
* Food journal are handed out - food intake over three consecutive days will be registered by the patient.

VISIT 2

* Handing in urine - the last of the urine collected on visit 1 is being handed in by the patient.
* Returning EKG-material - the Holter, recording EKG, is returned by the patient.

VISIT 3

* Salivary sample - test to measure the levels of cortisol, an important stress marker.
* Oro-anal transit time - 60 markers that can be seen through x-ray examination are being swallowed prior to the visit (10 markers/day during 6 days) and in the examination it is possible to see how many of the markers remain in the GI-tract and where in the tract they are positioned. This is a way to measure the oro-anal transit time, which mainly is determined by the colonic transit time. Thereby this is an indirect measurement of the motor function in colon. Regional transit in different colonic parts can be assessed by evaluating where in the colon the markers are.
* Rectal sensitivity testing - a balloon is placed in the rectum and is through a tube attached to a so called barostat. By using the barostat it is possible to inflate and deflate the balloon in a controlled matter and also to measure compression and volume in the balloon. The compression and volume is being increased in a predetermined way and the patient is asked to state how it feels by using VAS-scales; symptoms noted and the intensity of these symptoms. The sensitivity in the rectum (large intestine) can be described by valuing the levels of compression and volume that give rise to the symptoms.

VISIT 4

* Sigmoidoscopy with biopsies. Macroscopic evaluation of the mucosa of the large intestine, to rule out inflammatory bowel disease as a cause of the patients symptoms. Biopsies from the rectum and sigmoid are collected to be analyzed in regards of inflammatory cell populations and interleukins in the colonic mucosa, as well as amount of bacteria in the mucosa. Molecular techniques will be used, such as 16sRNA.
* Stool sample - analysis of immunological and inflammatory markers in the faeces and of the composition of the microbiological bacterial flora, this reflects the luminal bacterial flora (16sRNA technique will be used).
* Blood samples - various immunological analysis, for example different pro- and anti-inflammatory interleukins and different food related antibodies (IgE, IgG), are done to evaluate toe immunological activity and propensity to react in an unfavorable way when for instance consuming certain food items.
* Symptom protocol (IBS-SSS) and journal of stool consistency and frequency (Bristol Stool Form Scale (BSF)) are handed out. Symptoms and stools will be registered during 1-3 weeks and will be used as basal values prior to the treatment period.

VISIT 5

* Lactulose challenge test - evaluation of symptoms and excretion of hydrogen and methane gas in the exhaled air after intake of a liquid meal (400ml Nutridrink®, 1.5 kcal/ml) containing 25 mg lactulose. Hydrogen and methane gas in the exhaled air is a measurement of the degree of fermentation in the intestines, and indirectly can a bacterial overgrowth in the small intestine be detected. This "challenge" test is more of a physiological test to study the sensitivity of the GI-tract. The symptoms and excretion of gas will be registered during 4 h.
* Stool sample - analysis of immunological and inflammatory markers in the faeces and of the composition of the microbiological bacterial flora, this reflects the luminal bacterial flora (16sRNA technique will be used).
* Salivary sample - test to measure the levels of cortisol, an important stress marker.
* Randomization of the patients as they are included in the treatment part of the study. The patients will during 14 days have a daily intake of a yoghurt containing probiotics (Bifidobacterium lactis, Activia®) or a yoghurt without probiotics (placebo), 125 g 2 times a day (morning and evening). During the treatment part the patients register symptoms (Symptom protocol (IBS-SSS)) and stool consistency and frequency (Bristol Stool Form Scale (BSF)).

VISIT 6

* Visit takes place on the last day of the treatment period.
* Lactulose challenge test is being repeated to evaluate potential differences in symptoms and excretion of hydrogen and methane gas in the exhaled air after intake of a liquid meal (400ml Nutridrink®, 1.5 kcal/ml) containing 25 mg lactulose.
* Stool sample - analysis of immunological and inflammatory markers in the faeces and of the composition of the microbiological bacterial flora, this reflects the luminal bacterial flora (16sRNA technique will be used).
* Blood samples - various immunological analysis, for example different pro- and anti-inflammatory interleukins and different food related antibodies (IgE, IgG), are done to evaluate toe immunological activity and propensity to react in an unfavorable way when for instance consuming certain food items. Will be compared with previous blood samples.

VISIT 7

• Summarizing visit - visit at a doctor specialized in functional GI-disorders. The results from the tests and analysis of the previous visits are being evaluated and any potential treatment is based on these results. The patients are offered a telephone based follow-up if they want to, otherwise they are recommitted to the primary health care.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age: between 18 and 65 years old at baseline visit
* IBS according to the Rome III criteria
* Ability to understand and willingness to comply to the study procedures

Exclusion Criteria:

* Participation in another clinical study 1 month prior to screening visit and throughout the study
* Abnormal results on the screening laboratory tests clinically relevant for study participation
* Other gastrointestinal disease(s) explaining the patient's symptoms, as judged by the investigator
* Other severe disease(s) such as malignancy, severe heart disease, kidney disease or neurological disease
* Symptoms indicating other severe disease(s) such as gastrointestinal bleeding, weight loss or fever
* Severe psychiatric disease
* Previous history of drug or alcohol abuse 6 months prior to screening
* Intolerance or allergy against milk products or gluten
* Use of other probiotic products (according to sponsor's list) 2 weeks prior to the study and throughout the study
* Consumption of antibiotics 1 month prior to screening and throughout the study
* Consumption of cortisone, NSAID or other anti-inflammatory drugs on a regular basis 2 weeks prior to screening and throughout the study
* Pregnant or lactating or wish to become pregnant during the period of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
IBS symptoms | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Simrén, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg, Västra Götaland County
  - Dept of Internal Medicine, Sahlgrenska University Hospital, Gothenburg

REFERENCES:
- [Derived] Tap J, Storsrud S, Le Neve B, Cotillard A, Pons N, Dore J, Ohman L, Tornblom H, Derrien M, Simren M. Diet and gut microbiome interactions of relevance for symptoms in irritable bowel syndrome. Microbiome. 2021 Mar 26;9(1):74. doi: 10.1186/s40168-021-01018-9. PMID 33771219
- [Derived] Le Neve B, Derrien M, Tap J, Brazeilles R, Cools Portier S, Guyonnet D, Ohman L, Storsrud S, Tornblom H, Simren M. Fasting breath H2 and gut microbiota metabolic potential are associated with the response to a fermented milk product in irritable bowel syndrome. PLoS One. 2019 Apr 4;14(4):e0214273. doi: 10.1371/journal.pone.0214273. eCollection 2019. PMID 30946757
- [Derived] Nybacka S, Storsrud S, Liljebo T, Le Neve B, Tornblom H, Simren M, Winkvist A. Within- and Between-Subject Variation in Dietary Intake of Fermentable Oligo-, Di-, Monosaccharides, and Polyols Among Patients with Irritable Bowel Syndrome. Curr Dev Nutr. 2018 Dec 24;3(2):nzy101. doi: 10.1093/cdn/nzy101. eCollection 2019 Feb. PMID 30838348
- [Derived] Pohl D, Van Oudenhove L, Tornblom H, Le Neve B, Tack J, Simren M. Functional Dyspepsia and Severity of Psychologic Symptoms Associate With Postprandial Symptoms in Patients With Irritable Bowel Syndrome. Clin Gastroenterol Hepatol. 2018 Nov;16(11):1745-1753.e1. doi: 10.1016/j.cgh.2018.04.034. Epub 2018 Apr 24. PMID 29702295
- [Derived] Tap J, Derrien M, Tornblom H, Brazeilles R, Cools-Portier S, Dore J, Storsrud S, Le Neve B, Ohman L, Simren M. Identification of an Intestinal Microbiota Signature Associated With Severity of Irritable Bowel Syndrome. Gastroenterology. 2017 Jan;152(1):111-123.e8. doi: 10.1053/j.gastro.2016.09.049. Epub 2016 Oct 7. PMID 27725146
- [Derived] Le Neve B, Brazeilles R, Derrien M, Tap J, Guyonnet D, Ohman L, Tornblom H, Simren M. Lactulose Challenge Determines Visceral Sensitivity and Severity of Symptoms in Patients With Irritable Bowel Syndrome. Clin Gastroenterol Hepatol. 2016 Feb;14(2):226-33.e1-3. doi: 10.1016/j.cgh.2015.09.039. Epub 2015 Oct 20. PMID 26492847